CLINICAL TRIAL: NCT06872450
Title: Implementation and Impact Study of an Informational Tool for Smoking Cessation in COPD Patients
Brief Title: Informational Tool for Smoking Cessation in COPD Patients
Acronym: IMPACT-BPCO
Status: Completed | Type: Observational
Sponsor: Hopital Nord Franche-Comte (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-11-IMPACT BPCO
Record Dates: First submitted 2025-02-25; First posted 2025-03-12 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: informational and motivational tool
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- informational intervention: informational intervention
  Interventions: Other: informational intervention

INTERVENTIONS:
Other: informational intervention — informational intervention

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a lung disease that affects nearly 8% of the adult population and causes 18,000 deaths per year in France. The most frequent cause of this pathology is smoking. COPD patients who stop smoking have a better quality of life, a marked a significant slowdown in disease progression and an increased life expectancy. Investigators propose to carry out a quantitative study among patients smokers suffering from COPD, by setting up a tool in the form of an motivational intervention specific to this population.

DETAILED DESCRIPTION:
implementing a tool in the form of an informational intervention with a specific motivational intervention

ELIGIBILITY:
Inclusion Criteria:

* People suffering from chronic obstructive pulmonary disease (COPD) stage 2/3
* People treated at HNFC
* Smokers

Exclusion Criteria:

* People with cognitive disorders compromising comprehension and completion of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People suffering from chronic obstructive pulmonary disease (COPD) stage 2/3
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2025-02-14 (Actual); Primary Completion 2025-05-09 (Actual); Study Completion 2025-05-09 (Actual)

PRIMARY OUTCOMES:
motivational effectiveness | 60 days
  Motivation to stop smoking (QMAT test)
motivational effectiveness | 60 days
  Anxio-depressive state (HAD scale)
motivational effectiveness | 60 days
  Degree of dependence (Fagerström test)

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Nord Franche-comté, Trévenans, France

IPD SHARING:
Plan to Share IPD: No